CLINICAL TRIAL: NCT03874507
Title: Technology-Based Intervention for Physical Therapy in Pediatric and Adult Populations
Brief Title: Physical Therapy Using Virtual Reality/Augmented Reality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Thomas Caruso, Clinical Associate Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 50159
Record Dates: First submitted 2019-03-12; First posted 2019-03-14 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Mobility Limitation; Spinal Fusion; Acute Pain
Keywords: virtual reality; augmented reality; physical therapy; deconditioning
MeSH Terms: conditions — Mobility Limitation; Acute Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Technology-based therapy (Experimental): Patients who require acute rehabilitation due to deconditioning and surgery will receive either virtual reality (VR) or augmented reality (AR) to improve clinical outcomes such as range of motion, gait progression, strength progression, time to first out of bed, time to first step.
  Interventions: Other: Virtual Reality/Augmented Reality Headset
- Standard of Care therapy (No Intervention): Patients who require acute rehabilitation due to deconditioning and surgery will receive physical therapy based on his/her providers recommendations to improve outcomes such as range of motion, gait progression, strength progression, time to first out of bed, time to first step

INTERVENTIONS:
Other: Virtual Reality/Augmented Reality Headset — A virtual reality (VR) headset is a device the participant will wear over his/her head and eyes like a pair of goggles. It blocks out all external light and shows him/her an image on high-definition screens in front of his/hers eyes. It implies a complete immersion experience that shuts out the physical world.
  Augmented reality (AR) headset is a device that the participant will wear over his/hers head and eyes and it adds digital elements to a live view.
  Arms: Technology-based therapy

SUMMARY:
The purpose of this study is to determine if non-invasive distracting devices (Virtual Reality (VR) headset, Augmented Reality (AR) Headset) are more effective than the standard of care (i.e., no technology-based distraction) for improving clinical outcomes in patients requiring acute rehabilitation due to deconditioning and surgery. Measures will include include range of motion, gait progression, strength progression, time to first out of bed, time to first step.

ELIGIBILITY:
Inclusion Criteria:

* Age 6-99
* Diagnosis need for physical rehabilitation

Exclusion Criteria:

* Significant Cognitive Impairment
* History of Severe Motion Sickness
* Current Nausea
* Seizures
* Visual Problems
* Patients whose children are clinically unstable or require urgent/emergent intervention
* Patients who clinically unstable or requires urgent/emergent intervention

Ages: 6 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2019-07-25 (Actual); Primary Completion 2020-04-25 (Actual); Study Completion 2020-04-25 (Actual)

PRIMARY OUTCOMES:
Aggregate Movement | Duration of physical therapy, approximately 10 minutes
  Aggregate movement will be measured by either sensors in the VR/AR headset or by a physical therapist during the participants session
Patient and Physical Therapist Feedback | Survey of patient and PT satisfaction will be administered after the physical therapy session, duration of survey should take approximately 15 minutes or less
  Survey of patient and PT satisfaction will be administered after the session. Example of survey questions, to which patient answered 'Yes or No,' for patient include 1) 'The VR game helped me during physical therapy' 2) 'I felt less pain when I moved using the VR game' The survey administered to physical therapists will be rated 1-5 (1=Not at all, 5= A lot) with questions such as 1) 'The technology was helpful to my patients during physical therapy' and 2) 'I would like my patient to have access to this technology for future physical therapy sessions'
Patient Fatigue | OMNI PRE Questionnaire will be administered after the physical therapy session, duration of questionnaire should take approximately 15 minutes or less
  Patients will self-report fatigue according to the Adult OMNI-Walk/Run RPE Scale (OMNI RPE) scale after both the VR and standard of care portion. The OMNI RPE is an 11-category perceived exertion rating scale with a numerical rating from 0 to 10 (0= Not Tired at All, 10= Very, Very Tired).

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Lucile Packard Children's Hospital Stanford, Palo Alto, California
  - Stanford Health Care Hospital, Stanford, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hemphill S, Rodriguez S, Wang E, Koeppen K, Aitken-Young B, Jackson C, Simons L, Caruso TJ. Virtual Reality Augments Movement During Physical Therapy: A Pragmatic Randomized Trial. Am J Phys Med Rehabil. 2022 Mar 1;101(3):229-236. doi: 10.1097/PHM.0000000000001779. PMID 33935153